CLINICAL TRIAL: NCT03258086
Title: Assessment of Vitamin D in Children With Type 1 Diabetes
Brief Title: Vitamin D in Diabetic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17100043
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sample (Experimental): 2ml blood sample of of blood will be taken for assessment of vitamin D
  Interventions: Diagnostic Test: blood sample test

INTERVENTIONS:
Diagnostic Test: blood sample test — blood sample will be taken from all diabetic children for assessment of vitamin D level

SUMMARY:
Vitamin D is so-called "sunshine vitamin",it is synthesized in the skin during exposure to the ultraviolet rays in sunlight so it has been suggested that ∼ 5-30 minutes of sun exposure between 10:00 a.m. and 3:00 p.m. at least twice per week on the skin of the face, arms, back, or legs (without sunscreen) is usually adequate for vitamin D synthesis. Vitamin D is also found in plants (mainly mushrooms and yeast) and in a few foods such as fatty fish.

Vitamin D supplement is recommended in all infants until enough formula, milk, or other food sources are ingested to sufficiently provide 400 IU/day to prevent vitamin D deficiency. Type 1 diabetes is an autoimmune disease, and the self immune system plays a central role in the destruction of the beta cell of pancrease.

ELIGIBILITY:
Inclusion Criteria:

* Age (5 years - 15 years ).
* Type 1 diabetes patients.

Exclusion Criteria:

* Patients aged more than 15 years, less than 2 years.
* Type 2 diabetes.
* Neonatal diabetes.
* Patients with any complications from diabetes.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Assessment of vitamin D level (ng/ml) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided